CLINICAL TRIAL: NCT04146077
Title: Active Surveillance Methodology for Low Risk Prostate Cancer
Brief Title: Active Surveillance for Low Risk Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Collaborators: Moscow Regional Research and Clinical Institute (MONIKI) (Other Government); Pirogov Russian National Research Medical University (Other)
Responsible Party: Principal Investigator, Dmitry Enikeev, MD, PhD, Deputy director for Research, Institute for Urology and Reproductive Health, I.M. Sechenov First Moscow State Medical University
Other Study IDs: Sechenov-AS-19
Record Dates: First submitted 2019-10-28; First posted 2019-10-31 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma
Keywords: prostate cancer; active surveillance; low oncological risk
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An active surveillance protocol for patients diagnosed low-risk prostate cancer will be held. We plan to use PSA (prostate-specific antigen) testing, DRE (digital rectal examination), TRUS (transrectal ultrasound), MRI (magnetic resonance imaging) and follow-up biopsies to monitor patients and detect cancer progression in time.

ELIGIBILITY:
Inclusion Criteria:

* prostate adenocarcinoma verified by at least 12 core biopsy
* patient must understand the sense of research, agree to participate and sign a form of agreement
* low oncological risk according to EAU (European Association of Urology) Guidelines: stage T1-T2a, PSA<10 ng/ml, ISUP (International Society of Urological Pathologists score)=1 (Gleason score 3+3=6)
* not more than 33% cores with adenocarcinoma

Exclusion Criteria:

* previous treatment of prostate cancer
* other prostatic malignant neoplasms
* other oncological diseases
* treatment with 5-alfa-reductase inhibitors
* patient's refuse to continue study
* patient's desire to begin treatment

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with low risk prostate cancer, who gave informed consent to undergo active surveillance and to participate in this study, and had no previous treatment of prostate cancer or surgery at the prostate.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
cancer progression | 5 years
  Number of patients who had one of the following signs of cancer progression: new lesion on DRE proved by biopsy, or histological upgrade on follow-up biopsy, or involvement of more than 33% cores on follow-up biopsy

SECONDARY OUTCOMES:
surgical treatment due to infravesical obstruction by BPH | 5 years
  Number of patients who underwent any treatment due to BPH: endoscopic procedures, or simple prostatectomy, or punction cystostomy

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Urology and Reproductive Health, Sechenov University., Moscow, Russia